CLINICAL TRIAL: NCT02863484
Title: Dissection of the Outer Layer of the Lateral Wall of the Cavernous Sinus Decreases Bleeding as Compared to Direct Tumor Attack in Middle Fossa Meningiomas: A Randomized Controlled Trial
Brief Title: Cavernous Sinus Dissection and Bleeding in Meningiomas
Acronym: OCS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Hegazy, Dr., Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-44-2016
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Meningiomas of the Middle Cranial Fossa
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional surgery intra-dural (Active Comparator): This arm will be surgically operated by direct attack of the tumour after opening the dura
  Interventions: Other: surgery
- Pealing surgery extra-dural (Experimental): This arm the pealing of the outer layer of the lateral wall of the cavernous sinus will be done before the dura is opened. After the pealing is completed, the middle meningeal artery will be divided at the foramen spinosum. Then, the dura will be opened and the tumour attacked.
  Interventions: Other: surgery

INTERVENTIONS:
Other: surgery — pealing of the outer layer of the cavernous sinus

SUMMARY:
The blood loss will be compared in middle fossa meningiomas which will receive pealing of the outer layer of the lateral wall of the cavernous sinus and those which will not revive pealing before the dura is opened

DETAILED DESCRIPTION:
Cases with middle fossa meningiomas will be randomised to one of two surgical techniques. The first technique will involve pealing of the outer layer of the lateral wall of the cavernous sinus before the dura is opened and the tumour attacked, and the second group of cases will be operated by a standard technique, where the tumour will be directly attacked with out pealing of the outer layer of the lateral wall of the cavernous sinus. Blood loss will be monitored in each case by calculating the amount of blood in the suction container and subtracting it from the amount of fluids used for irrigation during surgery. The number of cotton patties and dressings will be also counted with each case as well as the number of gauzes used. The pre-operative complete blood picture will be documented particularly the haemoglobin , hematocrits and others. The same lab data will be also monitored after surgery. The amount of blood transfusion required will also be calculated in each case.

ELIGIBILITY:
Inclusion Criteria:

* Meningiomas of the middle cranial fossa

Exclusion Criteria:

* Meningiomas outside the middle cranial fossa

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Amount of blood loss as estimated by cubic centimetres during surgery | three months

SECONDARY OUTCOMES:
Radically of surgery as estimated by post-operative tumour volume in cubic centimetres on post-operative MRI | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hegazy, MD, Principal Investigator — Professor of neurosurgery, faculty of medicine, Cairo University
Locations (1):
- Kasralainy medical college, Cairo University, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No